CLINICAL TRIAL: NCT06666530
Title: Quality of Life Related to the Care of Women Living With HIV During the Perinatal Period
Acronym: QUASOVIH
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231651; 2023-A02061-44 (Other: ID-RCB)
Record Dates: First submitted 2024-10-21; First posted 2024-10-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women living with HIV: women living with HIV during the perinatal period
  Interventions: Other: Questionary

INTERVENTIONS:
Other: Questionary — Three self-questionnaires, either completed independently or with assistance, will be administered at inclusion (between the first obstetric ultrasound and 28 weeks of amenorrhea), during the third trimester of pregnancy, and at 1 year postpartum

SUMMARY:
"The improvement of patient care by assessing the Quality of Life Related to Care (QLRC) in pregnant women living with HIV is of great importance for informing decision-making, resource allocation, and health policy formulation Prospective descriptive survey of women living with HIV followed for a pregnancy in the Infectious diseases department of Bichat-Claude Bernard Hospital, PARIS, France, between the first obstetric ultrasound and the 28th week of amenorrhea.

After recruitment during a follow-up consultation:

Information regarding the prenatal and perinatal management of HIV and the infant's outcomes up to 12 months will be collected retrospectively through the medical records.

Three self-questionnaires, either completed independently or with assistance, will be administered at inclusion (between the first obstetric ultrasound and 28 weeks of amenorrhea), during the third trimester of pregnancy, and at 1 year postpartum."

DETAILED DESCRIPTION:
"The latest report from the WHO shows that with 1.3 million (between 970,000 and 1.6 million) HIV-positive pregnant women worldwide in 2020, HIV continues to be a major global public health issue. In France, approximately 2 out of 1,000 pregnant women are infected with HIV, resulting in about 1,500 births per year over the past fifteen years. Although therapeutic advances have not yet led to a cure for the infection, they have increased life expectancy, improved the quality of life for people living with HIV, and reduced mother-to-child transmission during pregnancy, childbirth, and breastfeeding. Indeed, the very low transmission rate during replication has been completely eliminated.

The measurement of quality of life is increasingly used to complement the clinical or biological management of a disease, as it provides data to evaluate the quality of patient care, identify additional care needs, and assess the effectiveness of interventions. This approach enhances patient experience and satisfaction with treatment, in contrast to traditional management, which focuses on disease progression.

Generally, pregnant women report a lower health-related quality of life due to the impact of pregnancy on their physiological and mental health. In addition to limited physical activities in early pregnancy, most pregnant women are likely to experience nausea, vomiting, dizziness, depression, nervousness, and anxiety throughout their pregnancy. Compared to HIV-negative pregnant women, HIV-positive pregnant women may also have poorer physical health, a greater susceptibility to depression, and worse mental health. Factors such as education level, number of children, pregnancy symptoms, and occupation are key determinants of Health-Related Quality of Life (HRQoL) for pregnant women.

Consequently, improving patient care by assessing HRQoL in HIV-positive pregnant women is crucial for informing decision-making, resource allocation, and health policy formulation.

Through this project, we will explore the HRQoL of women living with HIV during the perinatal period under the care of the Infectious diseases department at Bichat-Claude Bernard Hospital, PARIS, FRANCE.

In 2022, the Infectious diseases department of Bichat-Claude Bernard Hospital cared for 5,242 people living with HIV, including 544 women of childbearing age (under 43 years). From January 1, 2005, to December 31, 2022, 1,158 women living with HIV were monitored for pregnancy, with 1,036 delivering at Bichat-Claude Bernard Maternity.

During the period from January 1 to December 31, 2022, 43 women living with HIV were followed at Bichat Maternity during their pregnancy, and 38 gave birth to live infants at the hospital. Among these 38 women, the median age was 36 years (range: 20-50), and 86.8% were originally from Sub-Saharan Africa.

According to the report from the Interministerial Mission on Poverty and Social Exclusion, areas with the highest prevalence of poverty and social exclusion are located in the northern part of Paris and Île-de-France, and the Bichat-Claude Bernard hospital group is at the heart of this area. The PréCARE cohort study (which monitored pregnant women from October 2010 to May 2012) highlighted specific vulnerabilities in this territory, particularly among undocumented migrants who faced a higher risk of obstetric complications compared to women born in France.

The outpatient follow-up for pregnant women living with HIV has been designed to provide comprehensive health management during pregnancy, focusing not only on complications related to the infection or pregnancy but also on ensuring ""a state of complete physical, mental, and social well-being"" (WHO definition of health).

This approach ensures:

* Adherence to and good tolerance of antiretroviral therapy, as well as effective virological control of HIV infection
* Proper management of pregnancy
* Physical and psychological well-being
* Addressing potential social issues."

ELIGIBILITY:
"Inclusion Criteria

* Woman living with HIV
* Age ≥ 18 years
* Pregnant - due date between the first obstetric ultrasound and 28 weeks of amenorrhea
* Information provided about the study and the right to refuse participation

Exclusion Criteria

* Refusal to participate in the study
* Non-French speaker"

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women living with HIV followed for a pregnancy in the SMIT of Bichat-Claude Bernard Hospital, PARIS, France, between the first obstetric ultrasound and the 28th week of amenorrhea
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Collection of perceptions of pregnancy care via the Hospital Anxiety and Depression Scale | during the Perinatal Period at 1 Year Postpartum

SECONDARY OUTCOMES:
Describe the sociodemographic characteristics of the mothers | up to 1 year postpartum
Describe the course of pregnancy period through different parameters: HIV discovery setting, type of mother's income, administrative status, mother treatments, immunovirological control, intrapartum AZT infusion | up to 9 month
Describe the course of the postpartum period through different parameters: type of mother's income, administrative status, mother and child treatments, immunovirological control, delivery method, characteristics of newborns at birth | at 1 year postpartum
Describe the care of children born to women living with HIV : Collection of clinical and epidemiological data from children | up to 1 year
Describe the serological status of children born to women living with HIV (HIV+ or HIV-) | at 1 year
Describe the sharing of HIV status with the partner during pregnancy: yes or no and the reason for not sharing | up to 1 year postpartum
Collection of perceptions of pregnancy care | at 1 year postpartum
  personnal scale: feel good, feel "overwhelmed", feel reassured by the team that takes care of you, find this PEC too medicalized, which does not allow to fully enjoy pregnancy, find this PEC time-consuming and heavy and the reason
Describe the mother's perception of the care of the newborn | at 1 year postpartum
  personnal scale: reassures you, Worries you, Weighs you, You find it difficult to perform
Describe the mother's perception of the possibility of breastfeeding and conditions associated with breastfeeding | up to 1 year postpartum
  personnal scale: How do you feel about the contraindication to breastfeeding?
  I am happy; I am reassured; I am sad; I am angry; Others, specify:
Describe the evolution of the mother's anxiety and depression | up to 1 year postpartum
  Hospital Anxiety and Depression Scale
Describe the perception of the management of the previous pregnancy | 1 day
  personnal scale: You felt good; You felt "overwhelmed"; You felt reassured by the team taking care of you; You found this PEC too medicalized, which did not allow you to fully enjoy your pregnancy; You found this PEC time-consuming and heavy, specify why; You could not follow up properly, specify
Describe the reasons for non-inclusions: Patient refusal, Doctor refusal; Term pregnancy after 28 weeks; Does not speak French; Doesn't have time; Other | 1 day
describe breastfeeding practices | up to one year
  Duration, difficulties encountered, adherence to follow-up, and satisfaction
Describe maternal virological conditions associated with breastfeeding | up to one year
  maternal viral load during breastfeeding
describe pediatric conditions associated with breastfeeding | up to one year
  childhood prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Bachelard Antoine, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bichat-Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided